CLINICAL TRIAL: NCT02902731
Title: Randomized, Controlled, Double-blind Study of Anakinra Against Placebo in Addition to Steroids in Giant Cell Arteritis
Brief Title: Giant Cell Arteritis and Anakinra Trial
Acronym: GiAnT
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital, Caen (Other)
Collaborators: Hôpital Claude-Huriez (Other); Amiens University Hospital (Other); University Hospital, Rouen (Other); University Hospital, Limoges (Other); Central Hospital Saint Quentin (Other Government); Valenciennes Hospital, Valenciennes, FRANCE (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2015-005804-27 N° CHU : 15-200
Record Dates: First submitted 2016-07-05; First posted 2016-09-16 (Estimated); Last update posted 2020-02-25 (Actual); Status verified 2020-02

CONDITIONS: Giant Cell Arteritis
MeSH Terms: conditions — Giant Cell Arteritis | interventions — Interleukin 1 Receptor Antagonist Protein

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- placebo (Placebo Comparator): PLACEBO + Usual use of tapering doses of oral prednisone
  Interventions: Drug: PLACEBO
- anakinra (Experimental): ANAKINRA : dose of anakinra is 100 mg/day by subcutaneous injection from day 1 until the end of week 16 (W16). The dose of Anakinra will be adapted to that recommand according to renal function.
  Intervention Anakinra in add on Therapy.
  Interventions: Drug: ANAKINRA

INTERVENTIONS:
Drug: PLACEBO — subcutaneous injection of placebo every day during 16 weeks
  Other Names: comparative drug
  Arms: placebo
Drug: ANAKINRA — subcutaneous injection of anakinra every day during 16 weeks
  Arms: anakinra

SUMMARY:
SYNOPSIS The giant cell arteritis (GCA) is the most frequent vasculitis in people over 50 years. Despite recent progress and physiopathogenic, corticosteroids remains the standard treatment for decades with a very good initial clinical efficacy but a high relapse rate (nearly 40% to 6,5 months) during its decay. This sensible population is particularly exposed to the side effects of corticosteroids, leading to think about savings strategies. But the association of immunosuppressive therapy and/or anti- TNFα has not demonstrated benefits in terms of efficiency or long-term tolerance to cumulative doses of prednisone. The responsibility of proinflammatory cytokines such as TNFα, IL- 6 and IL-1 has been studied in the pathogenesis of GCA in temporal artery walls and in mouse models. The primary pathogenic role of IL- 1 is based on the increase in serum or nuclear protein itself or that of its mRNA. The study of temporal artery biopsies has shown increased local production of IL- 1β mRNA, IL- 6 and TGFβ (indicative of macrophage activation ) and those of INFɣ and IL 2 (indicative of T lymphocyte activation). Recently, Ly et al (Ly KH JBS 2014) reported the efficacy of anakinra, a recombinant molecule of IL- 1RA specifically blocking the IL- 1 α/β, in three cases GCA refractory to conventional treatments.

Here investigators propose a randomized, multicenter, controlled, double-blind study of anakinra against placebo in addition to corticosteroids in the treatment of GCA.

This study will include 70 patients randomized equally in both arms: reference treatment (prednisone plus placebo) or the experimental treatment (prednisone + anakinra). Treatment with prednisone will be identical in the two arms, namely a dose of 0.7 mg/kg/day orally on day 1, followed by a progressive decrease in the dose pattern depending on the weight. In the experimental arm, dose of anakinra is the one usually used, ie 100 mg/day by subcutaneous injection from day 1 until the end of week 16 (S16). In the reference arm of the treatment, a placebo anakinra is associated with corticosteroid in the same packaging, duration and respecting the double-blind.

Investigators thus hypothesized that the addition of anakinra to corticosteroid compared to placebo added to the latter, will show a significant decrease in GAC relapse rate. Indeed, the challenge of corticosteroid therapy in this disease is not so much a problem of initial effectiveness, than the adverse events related to relapses and steroid dependence.

DETAILED DESCRIPTION:
Side assumptions investigators made are that the patients receiving anakinra in add-on therapy will have: a time and a complete remission rate respectively shorter and higher, fewer relapses and a decrease of the total consumption of prednisone over a 12- month follow-up.

This controlled study is the first to assess the inhibition of the IL- 1 pathway in the GCA with anakinra in add-on therapy with corticosteroids in patients newly diagnosed or on relapse. The purpose of this work is to support the following proof of concept of the addition of anakinra to corticosteroid therapy in the treatment of GCA: potential synergies of this association and intrinsic therapeutic action of anakinra in patient newly diagnosed, and this without loss of opportunity for patients that will benefit all of the reference treatment. The other originality of this study is to demonstrate the steroid-sparing effect of targeting interleukin -1, which is per se a therapeutic and nosologic innovation for this disease. Finally, ancillary biological studies will clarify the mode of action of the anti-cytokine therapy and identify markers of response to this biotherapy.

ELIGIBILITY:
Minimum Age: 51 Years

Maximum Age:

Gender: Both Accepts Healthy Volunteers?: No

Criteria:

Inclusion Criteria: (Giant cell arteritis = GCA)

Age ≥ 50 years

Patient with temporal arteritis giant cell match 3 of the 5 criteria of the American College of Rheumatology (ACR) that:

Given a temporal artery biopsy compatible with a diagnosis of GCA (not necrotizing arteritis, giant cell with a granulomatous inflammatory infiltrate, usually localized to the intima-media junction, makes lymphocytes, macrophages and multinucleated giant cells; or minimum detection of a chronic inflammatory infiltrate fact lymphocytes and some neutrophils or eosinophils without giant cells).

Either abdominal thoracic aortitis diagnosed by:

* Angio CT: circumferential thickening of the aortic wall more than 3 mm, in the absence of adjacent plaque and active infection.
* MR angiography: wall thickening of the aortic wall with hyperintense on T1 weighted and T2 weighted enhancement after gadolinium injection.
* PET scanner: increased uptake of FDG by the aorta and its branches is not typical for GCA and may be in the atheroma. The PET scanner is probably a very sensitive technique but not specific enough to retain the diagnosis of GCA. We therefore consider the PET CT as a diagnostic method of secondary aortite the GCA if there simultaneously on the same exam fixing aortic (thoracic or abdominal) and blood of large caliber (artery (s) axillary ( s), subclavian (s) and / or carotid (s) of FDG.

Newly diagnosed disease and from corticosteroid started up to 14 days, the initial dose is less or equal to1 mg / Kg or

GCA recurrence of continuous therapy with corticosteroids (including hydroprednisone) and / or immunosuppression was stopped for at least 6 months. At the time of recurrence, at least 3 of 5 ACR criteria for the diagnosis of GCA must be present. Furthermore :

* if BAT (Biopsy of the temporal artery) was positive at the time of initial diagnosis, it is not necessary to make a new.
* if BAT was negative, the patient can not be included after completion of a new BAT which will be positive or if there is a aortite, evidenced by angio-CT or MR angiography or PET scanner.

For men and women of childbearing age, effective contraception must be used in the patient or his partner for the duration of treatment with anakinra (or placebo) and for 3 months after treatment. Also, breastfeeding is allowed after 3 months of stopping anakinra. Women considered not at risk of pregnancy are defined with menopause for at least a year or surgically sterile (tubal ligation, bilateral oophorectomy or hysterectomy)

Patient wo has given its written consent Patient affiliated with a social security

Exclusion Criteria:

Subjects checking one of the criteria for non-inclusion may be eligible to participate in the research. These criteria may include:

1. pathologies, habitus or other patient characteristics

   * Pregnancy, breastfeeding women or women of childbearing potential not using contraception
   * dementia syndrome
   * Patient not observing
   * Patients who live more than 150 km from the investigation center
   * ethyl or drug intoxication history that required hospitalization in the previous year
   * Patient monitoring and / or treated to another autoimmune disease or known inflammatory
   * Hypersensitivity to anakinra or any of its excipients (Sodium citrate (E331), sodium chloride, disodium edetate (E385), polysorbate 80 (E433), sodium hydroxide (E524), water for injections, substrates of origin: Escherichia coli proteins)
   * Person under judicial protection, guardianship
   * Person deprived of liberty
   * Person not beneficiaries of the social security system
2. Other therapeutic

   - Patient has already started (or stopped there less than 6 months) in a protocol or not frame to its ACG or another disease, treatment with anti TNF-alpha, methotrexate, cyclosporine, cyclophosphamide, dapsone or bolus corticosteroids.
   * Patients on long-term glucocorticoid for another condition
   * Early treatment of CAG disease with a dose> 1 mg / kg whatever the duration
   * Immunization with live vaccines / mitigated during the 8 weeks
3. Infectious diseases

   * Chronic viral hepatitis (acute or) B or C
   * HIV Infection
   * Persistent infection or severe infection requiring hospitalization or treatment with IV antibiotics during the 30 days prior to inclusion
   * Infection requiring an oral antibiotic treatment in the preceding 14 days inclusion
   * History of active tuberculosis, histoplasmosis or listeriosis
   * latent TB Signs (based on a history of untreated contagion, an opacity of greater than 1 cm in diameter on chest x-ray, or an in vitro test (Quantiferon Gold or T-Spot TB) positive. A history of tuberculosis disease or latent TB whose treatment is completed and has been properly conducted is not an exclusion criterion, whatever the result of Quantiferon or T-Spot TB.
4. Unstable disease

   * Uncontrolled diabetes with a history of recurrent infections
   * unstable ischemic heart
   * Heart failure ≥ stage III / IV NYHA
   * Stroke recent (<6 months)
   * Or any other severe disease resulting in the opinion of the investigator, a risk to the patient due to its participation in the study.
5. A vascular risk, metabolic, infectious, neoplastic renal or as follows:

   • Patient at high cardiovascular risk: heart disease or vascular history of proven, type 2 diabetes at high cardiovascular risk *, vascular risk> 20% at 10 years (Framingham equation) Dyslipidemia • severe uncontrolled lipid-lowering therapy
   * Active Liver disease and liver failure
   * Neutropenia (<1500 / mm3) at the time of the introduction of Kineret / Placebo; and a patient with initial neutropenia may be included in the study if it corrects under Cortancyl®, and that the experimental treatment (Anakinra-Kineret / PLACEBO) may be commenced within 15 days after prednisone.

   Neoplasia under 5 years except carcinoma in situ of the cervix and skin cancer (excluding melanoma) with complete excision whose boundaries pass in safe area.

   • Severe renal impairment (clearance <30mL / min)

   * The high cardiovascular risk patients with diabetes are defined by:

   - A kidney disorder (proteinuria> 300mg / 24h or creatinine clearance <60mL / min according to Cockroft)

   - Or at least two of the following risk factors:

   - Men over 50 years, over 60 year old woman
   * History of premature coronary disease: myocardial infarction or sudden death in the father or relative in the first degree male before age 55 and before age 65 for females
   * Current or quit smoking for less than 3 years
   * High blood pressure treated or not
   * HDL cholesterol <0.40 g / L regardless of sex
   * Microalbuminuria (> 30 mg / 24h) NB: The moderate renal impairment (clearance ≥ 30 mL / min and <50 mL / min) is not here a criterion for non-inclusion, but the appropriate injection KINERET (anakinra) provided daily will be made every two days.

Min Age: 51 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2017-05-11 (Actual); Primary Completion 2020-03 (Estimated); Study Completion 2022-03 (Estimated)

PRIMARY OUTCOMES:
global relapse rate | Week 26

SECONDARY OUTCOMES:
specific relapse rate | Week 4 to Week 16
specific relapse rate | Week 17 to Week 26
specific relapse rate | W27 to W52
speed efficiency : time of obtaining a complete remission over a follow up of 52 weeks period | baseline up to 52 weeks
number of first relapse | baseline up to 52 weeks
cumulative and the average dose of prednisone used | baseline up to 52 weeks
Safety according CTCAE v4.0 | baseline up to 52 weeks

OTHER OUTCOMES:
T-cells (Th1, Th2, Th17 et Treg) et T CD8 (Tc1, Tc2, Tc17) | at Week 0, Week 16
Cytokines (IL-6, IL-17, IFN-γ, IL-1β et TNF-α) | at Week 0, Week 16
  1. T-cells (Th1, Th2, Th17 et Treg) et T CD8 (Tc1, Tc2, Tc17)
  2. Cytokines (IL-6, IL-17, IFN-γ, IL-1β et TNF-α)
  3. vascular smooth muscles, fibroblastes (cytokines, inflammasome)
vascular smooth muscles, fibroblastes (cytokines, inflammasome) | at Week 0, Week 16

CONTACTS AND LOCATIONS:
Overall Officials: Achille AOUBA, MD PHD, Principal Investigator — CHU CAEN
Locations (1):
- Pr Aouba, Caen, France

IPD SHARING:
Plan to Share IPD: Undecided
It will be planify

REFERENCES:
- [Derived] de Boysson H, Ly KH, Geffray L, Quemeneur T, Liozon E, Bezanahary H, Gouellec NL, Audemard A, Dumont A, Deshayes S, Boutemy J, Maigne G, Martin Silva N, Sultan A, Le Mauff B, Petit G, Parienti JJ, Aouba A. Four months of treatment with anakinra combined with glucocorticoids for giant cell arteritis: a multicenter, randomized, double-blind, placebo-controlled trial. Arthritis Res Ther. 2025 Jun 7;27(1):122. doi: 10.1186/s13075-025-03493-z. PMID 40483523
- [Derived] Sun MM, Pope JE. Polymyalgia rheumatica and giant cell arteritis: diagnosis and management. Curr Opin Rheumatol. 2025 Jan 1;37(1):32-38. doi: 10.1097/BOR.0000000000001059. Epub 2024 Oct 14. PMID 39400109